CLINICAL TRIAL: NCT06486207
Title: Effects of Kendall Exercise VS Gong's Mobilization on Pain, Range of Motion, Function, and Strength in Cases With Upper Cross Syndrome
Brief Title: Effects of Kendall Exercise VS Gong's Mobilization on Pain, Range of Motion, Function, and Strength in Cases With UCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/727
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Syndrome, Down
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong's mobilization (Experimental)
  Interventions: Combination Product: Gong's mobilization
- Kendall Exercise (Other)
  Interventions: Other: Kendall Exercise

INTERVENTIONS:
Combination Product: Gong's mobilization — increases the range of motion for shoulder medial rotation by allowing shoulder medial rotation with the humeral head in a normal position against the glenoid cavity of the scapula
  Arms: Gong's mobilization
Other: Kendall Exercise — The Kendall exercise methods were as follows: Strengthening the deep cervical flexors, lying flat on the back with the chin down and then lifting the head and holding this position for 2-8 seconds to strengthen deep cervical flexors
  Arms: Kendall Exercise

SUMMARY:
The effectiveness of kendall exercise vs. gong's mobilization for alleviating pain with improvment in range of motion, function and strength in cases with upper cross syndrome, assessed by dividing 44 patinets in two groups as Group A (n=22) was treated with Kendall exercises and Group B (n=22) managed by Gong's mobilization. VAS, NDI, SPADI, Goniometer and Dyanometer were used for assessing primary and secondary outcomes in patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45-65 years old
* Both genders
* Diagnosed with upper cross syndrome (UCS)
* Rounded shoulders
* Forward head posture
* Tightness in the pectoralis major and minor muscles 7. Weakness in the lower trapezius and rhomboid muscles
* Reporting neck pain, shoulder pain, or headaches

Exclusion Criteria:

* History of neck or shoulder surgery or trauma
* Presence of other musculoskeletal conditions affecting the cervical spine or shoulder girdle
* Inflammatory conditions such as rheumatoid arthritis or gout
* Neurological conditions affecting upper limb function
* Pregnancy
* Uncontrolled cardiovascular or respiratory conditions
* Contraindications to manual therapy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual Aanalogue scale | 12 Months
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.
Range of motion | 12 months
  Range of motion of cervical spian and shoudler joint measured using a goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Civil Hospital Khaniwal, Khānewāl, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No